CLINICAL TRIAL: NCT00524290
Title: Multinational Study of Acinetobacter Bloodstream Infection: Clinical Outcomes and Global Epidemiology-PITT Protocol
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Yohei Doi, Associate Professor, University of Pittsburgh
Other Study IDs: PRO07080043
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Acinetobacter Infections
Keywords: Acinetobacter; infection; isolate
MeSH Terms: conditions — Acinetobacter Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objectives of this multinational study are to assess the clinical outcomes of patients with Acinetobacter bloodstream infection and to further assess the predictors of mortality in this patient population. We also aim to characterize the molecular epidemiology of this remarkable organism in an attempt to further understand its transmission dynamics on a global level and to determine whether increased pathogenicity is geographically dependent.

DETAILED DESCRIPTION:
Medical records will be reviewed and information collected to assess the clinical outcomes of patients with Acinetobacter bloodstream infection and to further assess the predictors of mortality in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acinetobacter infections

Exclusion Criteria:

* Those that do not meet entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acinetobacter infections
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States